CLINICAL TRIAL: NCT04921436
Title: Modulation of Microbiota Metabolism in Cardiac Surgery Patients With at High Risk of Postoperative Multiple Organ Dysfunctions
Brief Title: Modulation of Microbiota Metabolism in Cardiac Surgery Patients
Acronym: MMMMODCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Petrovsky National Research Centre of Surgery (Other)
Collaborators: Federal Research and Clinical Centre of Intensive Care Medicine and Rehabilitology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 10031967MM
Record Dates: First submitted 2021-05-24; First posted 2021-06-10 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Multiple Organ Dysfunction
Keywords: microbiota;; sepsis;; antibiotics;; cardiac surgery
MeSH Terms: conditions — Sepsis | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Intervention Model Description: In group I, antibiotics-inhibitors of microbial metabolism are used in the perioperative period and the next 2 postoperative days The second group uses standard antibiotic prophylaxis
Who Masked: Participant
Masking Description: the first patient gets into the group of preventive therapy, the next one does not get into the group, and so on (1:1)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cardiac surgery patients with preventive treatment (Experimental): In addition to standard antibiotic prophylaxis (cefazolin 2 g 60 minutes before skin incision and 2 g 3 times a day after surgery), the following antibiotic regimens will be used perioperatively:
  Doxycycline (the day before surgery 200 mg and 100 mg on days 1 and 2 after surgery) or Rimfampicin (150 mg 2 times a day before and after surgery) + Gentamicin (240 mg 3 times a day before and 2 days after surgery) or Clarithromycin (500 mg once daily for up to 2 days after surgery).
  The route of administration (oral / intravenous) will depend on the condition of the patient.
  Interventions: Procedure: cardiac surgery
- cardiac surgery patients without preventive treatment (No Intervention): standard antibiotic prophylaxis (cefazolin 2 g 60 minutes before skin incision and 2 g 3 times a day after surgery)

INTERVENTIONS:
Procedure: cardiac surgery — prophylactic use of antibiotic-inhibitors
  Arms: cardiac surgery patients with preventive treatment

SUMMARY:
An imbalance in the microbiota (most often intestinal) largely determines the onset of a disease state, and often a critical state. Cardiac surgery accompanied by heart failure and hypoperfusion is a proven risk factor for the development of metabolic disorders of the intestinal flora and bacterial translocation. Previously, it was shown that the change in serum concentrations of phenolic metabolites of the intestinal microbiota reflects the dynamics of the severity of the patient's condition and can be used for objective monitoring of treatment. Preoperative analysis of microbial metabolites makes it possible to reliably identify the group of patients with the highest risk of developing postoperative organ dysfunctions. In patients with a baseline level of the sum of phenolic acid concentrations over 3.5 mmol / L, the likelihood of postoperative complications is 10 times higher (OR - 10.5; 95% CI 1.35-81.7, p = 0.026). Reducing the metabolic activity of opportunistic bacteria and the level of aromatic microbial metabolites associated with sepsis through the prophylactic use of antibiotics belonging to the group of protein synthesis inhibitors at the level of bacterial cell ribosomes is of great interest.

DETAILED DESCRIPTION:
MMMMODCS (Modulation of Microbiota Metabolism Multiple Organ Dysfunctions in Cardiac Surgery) is a single-center clinical study, during which it is planned to study the safety and efficacy of the perioperative use of antibiotic inhibitors of protein synthesis at the ribosome level of bacterial cells (hereinafter: antibiotic inhibitors) in patients with the high risk of developing multiple organ dysfunction (MOD) of infectious genesis. The high-risk group is represented by patients who are planned to have surgery on the thoracoabdominal aorta; combined operations on coronary vessels and heart valves; patients with initially low heart ejection fraction (less than 45%). The study was designed to find out if the prophylactic use of a combination of antibiotic inhibitors prevents an increase in concentration (or contributes to a decrease with an initial increase) of aromatic microbial metabolites (AMM) above 3.5 mmol / L and the development of MOD, requiring a long stay in the intensive care unit more than 6 days). After signing an informed consent prior to surgery, patients will be randomized into one of two cohorts: with or without a combination of antibiotic inhibitors.

In a cohort with prophylactic treatment, in addition to standard antibiotic prophylaxis (I, II generation cephalosporins), combinations of the following antibiotic inhibitors (Doxycycline or Rimfampicin + Gentamicin or Clarithromycin) will be used orally or intravenously, depending on the patient's condition.

The AMM level will be measured in blood serum samples on a gas chromatography-mass spectrometer before the operation, on the 3rd and 6th days after the operation. The rest of the indicators will be discussed at the same points.

ELIGIBILITY:
Inclusion criteria:

* patients with aneurysmal aortic disease / aortic rupture;
* patients with ischemic heart disease and dysfunction of the valves;
* patients with initially low heart ejection fraction (less than 45%).

Exclusion criterion:

* tolerance to antibacterial drugs;
* taking oncological chemotherapy drugs;
* taking probiotics and nutritional supplements within the last month;
* intraoperative complications (shock of any etiology, allergic reactions).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-03 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
AMM level | 3 - 6 days after surgery
  the frequency of detecting patients with an AMM level in the blood serum of no more than 3.5 μmol / l (according to the results of GC-MS analysis)
the duration of stay in the ICU | one week
  the frequency of detecting patients

SECONDARY OUTCOMES:
adverse events associated with taking antibiotics (allergic / anaphylactic reactions); cases of sepsis (according to the criteria of Sepsis-3) / septic shock; patients with SOFA more than 7 points more | 6 days after surgery
  the frequency of detecting patients

CONTACTS AND LOCATIONS:
Overall Officials: MAXIM BABAEV, D.Sc., Principal Investigator — Petrovsky National Research Centre of Surgery
Locations (1):
- Petrovsky National Reasearch Centre of Surgery, Moscow, Russia